CLINICAL TRIAL: NCT02312271
Title: Enteral Formula Tolerance of Standard Tube Feedings
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 14.01.US.HCN
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Enteral Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- enterally fed adults: adult subjects with established enteral access receiving standard tube feeding formula
  Interventions: Other: enteral formula

INTERVENTIONS:
Other: enteral formula — standard tube feeding formulas

SUMMARY:
This prospective observational study seeks to assess ability to achieve enteral feeding goals with standard tube feeding formulas.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Currently tolerating enteral feeding
* Has enteral access
* Requires enteral tube feeding to provide 90% or more of their nutritional needs (without the use of modular(s)) for at least 21 days
* Having obtained his/her and/or his/her legal representative's informed consent.

Exclusion Criteria:

* Condition which contraindicates enteral feeding (i.e. intestinal obstruction)
* Lack of enteral access
* Any condition that would contraindicate use of the study product (i.e. need for severe fluid restriction, cow's milk protein allergy, other)
* Currently participating in another conflicting clinical study that would interfere with anticipated endpoints
* Judged to be at risk for poor compliance to the study protocol.
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with established enteral access receiving standard tube feeding formula
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Daily percentage of caloric nutritional goal met | 21 days

SECONDARY OUTCOMES:
Daily percentage of protein goal met | 21 days
GI tolerance | 21 days
Adverse events and serious adverse events | 21 days

CONTACTS AND LOCATIONS:
Locations (3):
- United States (2):
  - University of Arkansas, Little Rock, Arkansas
  - Vanderbilt University, Nashville, Tennessee
- Bruyere Research Institute, Ottawa, Ontario, Canada